CLINICAL TRIAL: NCT06363565
Title: Study on the Effect of Compound Nutrients on Reducing Homocysteine -- A 3-month Double-blind Randomized Controlled Trial
Brief Title: Effects of Supplementation of Compound Nutrients on Plasma Homocysteine in Chinese Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huilian Zhu, Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MN-2022-11
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Homocysteine
MeSH Terms: interventions — Folic Acid; Vitamin B 6; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supplementation of compound nutrients (Experimental): Folic acid, vitamin B6, vitamin B12, and betaine are provided as a 1.0g tablet. the tablet is orally taken twice a day, two tablets at a time 12 weeks.
  Interventions: Dietary Supplement: supplementation of compound nutrients
- placebo control (Placebo Comparator): The placebo is an excipient and the color, flavor, shape, taste, and weight are same with the tablet of folic acid, vitamin B6, vitamin B12, and betaine supplement.
  Interventions: Dietary Supplement: placebo control

INTERVENTIONS:
Dietary Supplement: supplementation of compound nutrients — Folic acid, vitamin B6, vitamin B12, and betaine per day orally for 12 weeks.
  Other Names: Folic acid, vitamin B6, vitamin B12, and betaine supplement
  Arms: supplementation of compound nutrients
Dietary Supplement: placebo control — The placebo is an excipient and the color, flavor, shape, taste, and weight are same with the tablet of supplement.
  Arms: placebo control

SUMMARY:
The purpose of this study is to determine whether supplementation of compound nutrients, including folic acid, vitamin B6, vitamin B12, and betaine, will decrease the level of plasma homocysteine in Chinese adults with homocysteine levels above 10 μmol/L.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 - 65 years;
2. Concentration of plasma homocysteine is between 10 and 100 μmol/L;
3. Free from any supplements or drugs that may decrease plasma homocysteine concentration for at least 1 month prior to the beginning of study;
4. Willing to participate in the study and sign informed consent.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Allergic physique or allergic to our compound nutrients tablets;
3. Complicated with severe diseases;
4. Unable to conduct study procedures;
5. Participating in any other intervention studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
levels of homocysteine | 12 weeks
  At baseline, 4 weeks, and 12 weeks, blood samples will be drawn and levels of homocysteine will be determined in the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Huilian Zhu, professor, Study Chair — Sun Yat-sen University
Locations (1):
- SunYat-sen University, Guangzhou, Guangdong, China